CLINICAL TRIAL: NCT00097006
Title: Retrovirus Epidemiology Donor Study-II (REDS-II)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1243
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2009-09

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Donors; Blood Transfusion; HIV Infections; HIV-1; HIV-2; HTLV-I; HTLV-II; Retroviridae Infections; Hepatitis, Viral, Human; Hepatitis B; Hepacivirus; West Nile Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Retroviridae Infections; Hepatitis, Viral, Human; Hepatitis B

SUMMARY:
To conduct epidemiological, laboratory, and survey research on volunteer blood donors within the United States to ensure the safety and availability of the United States' blood supply.

DETAILED DESCRIPTION:
BACKGROUND:

REDS-I was established to address important blood safety issues involving human retroviruses. On July 17, 1989 the NHLBI awarded contracts to five major blood centers and a coordinating center to develop a major multicenter epidemiologic study of the human retroviruses HIV-1, HIV-2, HTLV-I, and HTLV-II in volunteer U.S. blood donors. The original mission of REDS-I was to initiate and facilitate investigations of human retroviruses in volunteer blood donors from areas of the country at varying risk for HIV. During the course of the project, NHLBI expanded the original REDS-I mission to investigate critical questions posed by the blood banking and transfusion medicine communities that were essential to ensuring an adequate blood supply without compromising blood safety. The overall REDS-I program includes epidemiologic, laboratory, and clinical investigations, and provides a comprehensive framework for monitoring U.S. blood donations, and more recently transfusion recipients, for infectious disease markers. The operational and database structure of REDS-I, specifically designed to study U.S. blood safety and availability, has also provided a framework for rapid analytical response to other research questions of significant importance to the safety of the blood supply. Since its inception, investigators have made major contributions in assessing: the risk of contracting transfusion-transmitted infectious agents; HIV and HCV test screening; donor characteristics and behaviors; and ways of reducing HIV risk from transfusion. REDS-I investigators work closely with the Food and Drug Administration (FDA), Centers for Disease Control and Prevention (CDC) and Office of the Secretary, Department of Health and Human Services (DHHS) to provide data and analyses for important policy decisions. Liaisons with test manufacturers have enabled the rapid study of test procedures of critical importance to blood safety and availability.

DESIGN NARRATIVE:

The objectives of the Retrovirus Epidemiology Donor Study-II (REDS-II) are to conduct epidemiological, laboratory, and survey research on volunteer blood donors within the United States to ensure the safety and availability of the United States' blood supply. This includes monitoring known blood-borne infectious agents, rapidly evaluating the impact of emerging pathogens, assessing the safety implications of changes in laboratory and/or blood donor screening protocols and examining blood supply and availability issues. Addressing issues concerned with the safety and availability of the United States' blood supply will be the cornerstone of the National Heart, Lung, and Blood Institute's Retrovirus Epidemiology Donor Study. These issues include: a) the risks of transfusion-transmissible infections and their trends through time--these include infectious agents currently undergoing laboratory screening as well as new and emerging agents such as West Nile Virus (WNV) which is about to be screened for in the U.S. under experimental protocols; b) ways to reduce the risks of transfusion-transmissible infections; c) HIV, HTLV, HCV, and HBV test screening methodologies; d) donor characteristics, behaviors, and donation return patterns of U.S. blood donors; and e) the effectiveness and safety of various strategies implemented to increase the U.S. blood supply.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Busch — Vitalant Research Institute; Jerome Gottschall — Blood Center of Southeastern Wisconsin, Inc.; Christopher Hillyer — Emory University; Ram Kakaiya — Institute for Transfusion Medicine; Edward Murphy — University of California, San Francisco; Jorge Rios — American Red Cross Blood Services, New England Region; Ronald Sacher — University of Cincinnati; George Schreiber — Westat, Inc.

REFERENCES:
- [Derived] Mast AE, Schlumpf KS, Wright DJ, Johnson B, Glynn SA, Busch MP, Olbina G, Westerman M, Nemeth E, Ganz T; NHLBI Retrovirus Epidemiology Donor Study-II (REDS-II). Hepcidin level predicts hemoglobin concentration in individuals undergoing repeated phlebotomy. Haematologica. 2013 Aug;98(8):1324-30. doi: 10.3324/haematol.2012.070979. Epub 2013 Feb 26. PMID 23445875
- Available data/document: Individual Participant Data Set: REDS II-CORE — http://biolincc.nhlbi.nih.gov/studies/core/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Manual of Procedures: REDS II-CORE — http://biolincc.nhlbi.nih.gov/studies/core/
- Available data/document: Individual Participant Data Set: REDS II-LAPS — http://biolincc.nhlbi.nih.gov/studies/laps/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol: REDS II-LAPS — http://biolincc.nhlbi.nih.gov/studies/laps/
- Available data/document: Study Forms: REDS II-LAPS — http://biolincc.nhlbi.nih.gov/studies/laps/
- Available data/document: Manual of Procedures: REDS II-LAPS — http://biolincc.nhlbi.nih.gov/studies/laps/
- Available data/document: Individual Participant Data Set: REDS II-MS — http://biolincc.nhlbi.nih.gov/studies/redsms/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol: REDS II-MS — http://biolincc.nhlbi.nih.gov/studies/redsms/
- Available data/document: Manual of Procedures: REDS II-MS — http://biolincc.nhlbi.nih.gov/studies/redsms/
- Available data/document: Individual Participant Data Set: REDS II-RISE — http://biolincc.nhlbi.nih.gov/studies/rise/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol: REDS II-RISE — http://biolincc.nhlbi.nih.gov/studies/rise/
- Available data/document: Study Forms: REDS II-RISE — http://biolincc.nhlbi.nih.gov/studies/rise/
- Available data/document: Manual of Procedures: REDS II-RISE — http://biolincc.nhlbi.nih.gov/studies/rise/